CLINICAL TRIAL: NCT05538390
Title: Assesment of Pattern of Abdominal Injury Over a Two Year Period at St Paul's Hospital Millennium Medical College and AaBET Hospital, Addis Ababa, Ethiopia: A Retrospective Study
Brief Title: Assessment of Pattern of Abdominal Injury
Status: Completed | Type: Observational
Sponsor: St. Paul's Hospital Millennium Medical College, Ethiopia (Other)
Responsible Party: Sponsor
Other Study IDs: StPaulsHMMc
Record Dates: First submitted 2022-09-05; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Abdominal Trauma
Keywords: Abdominal Injury; Road traffic injury; Emergency department
MeSH Terms: conditions — Abdominal Injuries; Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other:

SUMMARY:
This hospital-based cross-sectional study was done at SPHMMC and AaBET hospitals from January 2018 to December 2019.The study aimed to assess the pattern of abdominal injury at St Paul's Hospital Millennium Medical College (SPHMMC) and Addis Ababa Burn, Emergency and Trauma (AaBET) hospital, Addis Ababa Ethiopia.Data was collected from the trauma registry and patient files using a pretested structured questionnaire filled out by two trained data collectors.The collected data was entered and analyzed using statistical software SPSS version 25.0.

DETAILED DESCRIPTION:
Data was collected from the trauma registry and patient files using a pretested structured questionnaire filled out by two trained data collectors. The questionnaire was categorized into socio-demographics (age, sex, residency, and address), clinical profile (triage, v/s, type of injury, associated injury), management, and outcome (management, complication, disposition, and mortality). Completeness of data was checked by the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

- All patients who are diagnosed clinically to have abdominal trauma

Exclusion Criteria:

* Patients who died before diagnosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients who presented to the AaBET and SPHMMC Hospital emergency department with a clinical diagnosis of abdominal trauma during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Pattern of Abdominal Injury | Over 2 years
  Frequency was analyzed in respective to socio-demographics (age, sex, residency, address), clinical profile(triage, v/s, type of injury, associated injury), management and outcome (management, complication, disposition and mortality) in patients presented with Abdominal injury in the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Kassaye D Altaye, Principal Investigator — University of Gondar
Locations (1):
- St Paul's Hospital Millennium Medical College, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: No
The data used to support the findings of this study are available from the Principal investigator upon request.

REFERENCES:
- [Result] Alastair, C.J., Pierre, J.G. Abdominal trauma. In: John M, Graeme D, Kevin OM, editors. Surgical Emergencies, 1st edition. Italy: Blackwell Science Ltd. 1999. 224-236
- [Result] Adesanya AA, Afolabi IR, da Rocha-Afodu JT. Civilian abdominal gunshot wounds in Lagos. J R Coll Surg Edinb. 1998 Aug;43(4):230-4. PMID 9735644
- [Result] Long MK, Vohra MK, Bonnette A, Parra PDV, Miller SK, Ayub E, Wang HE, Cardenas-Turanzas M, Gordon R, Ugalde IT, Allukian M, Smith HE. Focused assessment with sonography for trauma in predicting early surgical intervention in hemodynamically unstable children with blunt abdominal trauma. J Am Coll Emerg Physicians Open. 2022 Jan 27;3(1):e12650. doi: 10.1002/emp2.12650. eCollection 2022 Feb. PMID 35128532
- [Result] Abebe K, Bekele M, Tsehaye A, Lemmu B, Abebe E. Laparotomy for Abdominal Injury Indication & Outcome of patients at a Teaching Hospital in Addis Ababa, Ethiopia. Ethiop J Health Sci. 2019 Jul;29(4):503-512. doi: 10.4314/ejhs.v29i4.12. PMID 31447524
- [Result] Chalya PL, Mabula JB. Abdominal trauma experience over a two-year period at a tertiary hospital in north-western Tanzania: a prospective review of 396 cases. Tanzan J Health Res. 2013 Oct;15(4):230-9. PMID 26591698
- [Result] AdejumoAA,ThairuY,EgentiN.Profile of abdominal trauma in federal teaching hospital, Gombe, North-east, Nigeria: A cross sectional study. Int J Innov Med Health Sci 2015; 4: 41-5
- [Result] Bashah DT, Dachew BA, Tiruneh BT. Prevalence of injury and associated factors among patients visiting the Emergency Departments of Amhara Regional State Referral Hospitals, Ethiopia: a cross-sectional study. BMC Emerg Med. 2015 Aug 25;15:20. doi: 10.1186/s12873-015-0044-3. PMID 26302780